CLINICAL TRIAL: NCT04846387
Title: High-resolution Mapping of the Human Brainstem During Continence and Micturition: in Vivo Noninvasive 7 Tesla fMRI Study
Brief Title: Mapping of the Human Brainstem During Continence and Micturition: Noninvasive 7-T fMRI Study
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, Houston Methodist Hospital Urologist and Research Director, The Methodist Hospital Research Institute
Other Study IDs: PRO00026967
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Pontine Storage Center (PSC); Functional Magnetic Resonance Imaging (fMRI); Lower Urinary Tract Symptoms (LUTS); Pontine Micturition Center (PMC); Neuroimaging; Periaqueductal Gray (PAG); Micturition; Bladder; Incontinence; Overactive Bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Females with Normal Bladder Function: Diagnostic Tests: functional MRI and urodynamic studies.
  During screening, subject will be asked to come to their appointment with a full bladder. For the uroflow, they will urinate into a special funnel connected to a measuring instrument in a private bathroom followed by measuring Post void residual volume through PVR scanner. This is to ensure that they do not have any urological issue which can disqualify them from the study. At this visit, we will also instruct them about the urine voiding-holding task, our noninvasive fMRI paradigm, which the subjects will be performing during the fMRI portion of the study at visit 2. A 7-Tesla Siemens MAGNETOM scanner will be used. A urinary pouch will be used to collect the participant's urine while in the scanner.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Post-Void Residual; Diagnostic Test: Uroflowmetry; Behavioral: Questionaire - AUA Symptom Score
- Males with Normal Bladder Function: Diagnostic Tests: functional MRI and urodynamic studies.
  During screening, subject will be asked to come to their appointment with a full bladder. For the uroflow, they will urinate into a special funnel connected to a measuring instrument in a private bathroom followed by measuring Post void residual volume through PVR scanner. This is to ensure that they do not have any urological issue which can disqualify them from the study. At this visit, we will also instruct them about the urine voiding-holding task, our noninvasive fMRI paradigm, which the subjects will be performing during the fMRI portion of the study at visit 2. A 7-Tesla Siemens MAGNETOM scanner will be used. A condom catheter will be used to collect the participant's urine while in the scanner.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Post-Void Residual; Diagnostic Test: Uroflowmetry; Behavioral: Questionaire - AUA Symptom Score

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — A T1-weighted Anatomical Image, Diffusion Weighted Image, and functional MRI (fMRI) of "empty bladder" image will be obtained.
  Additionally, fMRI image during "full bladder" state and voiding/holding tasks will be obtained.
Diagnostic Test: Post-Void Residual — The patient's post-void residual is determined using a portable ultrasound machine after emptying the bladder just prior to entering the MRI scanner and immediately after the MRI scan.
  Other Names: PVR
Diagnostic Test: Uroflowmetry — Patients will urinate into a funnel connected to an electric flow meter to record urine flow rates in mililters per second. This is used as part of the screening process.
Behavioral: Questionaire - AUA Symptom Score — Subjects will fill out questionnaire asking about urinary symptoms. The range is 0-35.
  Other Names: AUASS

SUMMARY:
The lower urinary tract (bladder, bladder neck, urethra and urethral sphincter) has two functions: Storage (Continence) and voiding (micturition). Lower urinary tract dysfunction (LUTD) includes symptoms in the storage phase (such as urinary frequency, urgency, incontinence) or micturition phase (such as voiding dysfunction, hesitancy and urinary retention), or both. Proper urinary tract function is controlled by a complex network of peripheral and central nervous system. A delicate and complex switch exists between storage of urine and elimination of urine and in humans, the control over this switch is located in brain stem. Although significant research efforts have been utilized to understand supraspinal neural control of LUTs in humans, our understanding of the brainstem in humans is very limited, mainly due to the small size of nuclei.

The extensive involvement of the brainstem in LUTS control has urged us to look into a better way to investigate and identify the brainstem nuclei involved throughout the entire bladder cycle, especially in neurogenic patients. To our knowledge, there has been no published study using high-resolution MRI (7 Tesla) to study the role of brainstem specifically in LUT. Brainstem evaluation in regards to LUT function in a thorough and accurate manner using high-resolution techniques is of high priority for benign urology and National Institute of Health. The findings from this proposal will lay the foundation to study of brainstem control in the bladder cycle in neurogenic patients with high-resolution neuroimaging, and will be seminal research in the field.

The investigators hypothesize that Grey matter (blood-oxygen-level-dependent BOLD) signals and functional connectivity (FC) evaluation of the brainstem regions involved in continence and micturition are superior in 7T when compared to 3T in humans allowing assessment of the variations between men and women. Brainstem Regions of Interest (ROIs) include Pontine Storage Center (PSC) ("L region of the pons) and PAG are expected to be activated during the storage (continence) phase and Pontine Micturition Center (PMC) ("M" region of the pons) are expected to be activated during the voiding (micturition) phase.

DETAILED DESCRIPTION:
The current proposal will be the first 7-Tesla study evaluating brain and specifically brainstem control over LUT. The study will utilize a noninvasive functional MRI (fMRI) protocol that allows for evaluation of brainstem activity during continence and micturition in real-time, using high-resolution neuroimaging techniques (7T fMRI) in both men and women. The study will recruit 20 healthy subjects (10 male and 10 female) for participation in this study. The participants for this study will undergo a few tests including a uroflow, PVR and a protocol training session during screening at visit 1, and a fMRI at visit 2.

During screening, subject will be asked to come to their appointment with a full bladder. For the uroflow, they will urinate into a special funnel connected to a measuring instrument in a private bathroom followed by measuring Post void residual volume through PVR scanner. This is to ensure that they do not have any urological issue which can disqualify them from the study. At this visit, we will also instruct them about the urine voiding-holding task, our noninvasive fMRI paradigm which will involve having the participant drink 500-750 mL of water approximately 20 minutes prior to the start of their scan, which the subjects will be performing during the fMRI portion of the study at visit 2.

The subsequent Grey matter (BOLD) signals and functional connectivity (FC) analysis will allow investigators to further the current understanding of brainstem control of the LUT and bladder cycle.

ELIGIBILITY:
Inclusion Criteria:

• Healthy adult male and female volunteers ≥18 years of age with no neurological disease and genitourinary abnormalities will be screened:

* Post-Void Residual (PVR) < 20% of their bladder capacity OR
* Above 10 percentile of Liverpool nomogram

AND

• AUASS score < 7 will be eligible to participate in the study.

Exclusion Criteria:

* history of clinically relevant genitourinary malignancy or surgery such as:

  * anti-incontinence procedures
  * urethral strictures
  * advanced pelvic organ prolapse
* any neurological disorders
* history of seizures,
* pregnancy or planning to become pregnant,
* and contraindications to MRI will be excluded.
* Research team members who are involved with the data collection and the data analysis for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit healthy male and female volunteers > 18 years of age with no neurological disease and urinary issues at Houston Methodist Hospital.
  We anticipate an equal gender distribution (10 men and 10 women) among study participants.
  Once screened for inclusion and exclusion criteria, volunteers will be approached and asked if they would like to participate in this study. They will then be given study material and allowed sufficient time to make an informed decision regarding participation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signals intensity | 2 years
  BOLD signal intensity in the regions of interest during empty bladder, full bladder, and micturition in healthy males and females

SECONDARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signals | 2 years
  Differences in BOLD signal intensity in brainstem ROIs during micturition between genders
Uroflow measure | 2 years
  Maximum Qmax of urine (ml/sec): The range is between 0-40 mL/sec.
Postvoid Residual | 2 years
  Postvoid Residual (PVR) of urine in mL: The range is between 0-900 mL.
Urinary symptoms scores | 2 years
  Urinary symptom scores (no unit): The range is between 0-35. A higher score is associated with a worse outcome.
Mean Diffusivity (MD) | 2 years
  MD is a scalar value that describes the degree of diffusivity. MD of white matter tracts that are implicated in brain control of bladder are of interest.
Fractional Anisotropy (FA) | 2 years
  FA is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic (equally restricted) in all direction. No units. FA of white matter tracts that are implicated in brain control of bladder are of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States